CLINICAL TRIAL: NCT02629601
Title: Evaluating Incentive Designs to Increase Physical Activity Goal Adherence in a Wellness Program
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Change plans and no longer testing these interventions
Sponsor: University of Pennsylvania (Other)
Collaborators: Discovery Vitality (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 823617
Record Dates: First submitted 2015-12-07; First posted 2015-12-14 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Physical Activity
Keywords: physical activity; financial incentives; behavioral economics
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Active Rewards (Experimental): Participant will receive the standard active rewards incentives.
  Interventions: Behavioral: Active Rewards
- Active Rewards Doubled (Active Comparator): Participant will receive the standard active rewards doubled in magnitude.
  Interventions: Behavioral: Active Rewards Doubled
- Active Rewards & Lottery 1 (Active Comparator): Participant will receive the standard active rewards incentives plus a lottery 1 with a 1 in 3 chance of winning 3 times the reward and 1 in 100 chance of winning 40 times the reward.
  Interventions: Behavioral: Active Rewards; Behavioral: Lottery 1
- Active Rewards & Lottery 1 & Broadcast (Active Comparator): Participant will receive the standard active rewards incentives plus a lottery 1 with a 1 in 3 chance of winning 3 times the reward and 1 in 100 chance of winning 40 times the reward. Includes broadcasting winners (number) each week.
  Interventions: Behavioral: Active Rewards; Behavioral: Lottery 1; Behavioral: Broadcasting winners
- Active Rewards & Lottery 2 & Broadcast (Active Comparator): Participant will receive the standard active rewards incentives plus a lottery 2 with a 1 in 2 chance of winning 2 times the reward and 1 in 200 chance of winning 80 times the reward. Includes broadcasting winners (number) each week.
  Interventions: Behavioral: Active Rewards; Behavioral: Lottery 2; Behavioral: Broadcasting winners

INTERVENTIONS:
Behavioral: Active Rewards — Vitality standard active rewards wellness program for physical activity promotion
  Arms: Active Rewards; Active Rewards & Lottery 1; Active Rewards & Lottery 1 & Broadcast; Active Rewards & Lottery 2 & Broadcast
Behavioral: Lottery 1 — Participants have 1 in 3 chance of winning 3 times the reward and 1 in 100 chance of winning 40 times the reward
  Arms: Active Rewards & Lottery 1; Active Rewards & Lottery 1 & Broadcast
Behavioral: Lottery 2 — Participants have 1 in 2 chance of winning 2 times the reward and 1 in 200 chance of winning 80 times the reward
  Arms: Active Rewards & Lottery 2 & Broadcast
Behavioral: Broadcasting winners — Participants are told how many individuals won the lottery during that week.
  Arms: Active Rewards & Lottery 1 & Broadcast; Active Rewards & Lottery 2 & Broadcast
Behavioral: Active Rewards Doubled — Vitality standard active rewards wellness program for physical activity promotion with double the magnitude of incentives
  Arms: Active Rewards Doubled

SUMMARY:
This is a 4-week, five-arm, randomized, controlled trial to compare a standard wellness incentive program for physical activity to four other designs.

DETAILED DESCRIPTION:
Increased physical activity is associated with numerous health benefits including lower risk of cardiovascular disease. However, many individuals do not achieve physical activity goals. Vitality is a wellness program in South Africa that uses a program called "Active Rewards" to incentives achievement of weekly physical activity goals. In this study, the investigators will compare the standard active rewards program to doubling the magnitude or adding lottery designs with and without broadcasting the # of winners.

ELIGIBILITY:
Inclusion Criteria:

* Vitality member that has activated "active rewards" program

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Proportion of participants that acheived their weekly physical activity goal | 4 week intervention period
  Binary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Patel, MD, MBA, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No